CLINICAL TRIAL: NCT00348660
Title: The Seroprevalence of Hepatitis C and Course of Infection Among Pregnant Women Attending a Toronto Inner City Antenatal Care Clinic
Brief Title: Screening for Hepatitis C During Pregnancy at a Toronto Inner City Prenatal Clinic
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 04-095
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C; Pregnancy
Keywords: Screening for Hepatitis C in Pregnancy
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The first part of this study will investigate the incidence of Hepatitis C in pregnant women attending an inner city health clinic in downtown Toronto. All women attending the clinic who give their consent to participate will be screened by a standardized questionnaire as well as by a blood test. Blood testing will tell us how many of these women have Hepatitis C. We will then be able to compare the specificities and sensitivities of targeted screening (risk behaviour questionnaires) versus universal screening (blood tests).

In the second part of the study we will follow the pregnancies of those women who were identified as Hepatitis C positive on the screening test. Follow- up will include liver enzymes and viral load quantifications (amounts) in the first, second and third trimesters as well as during delivery and six weeks post-partum. We will also document pregnancy outcomes with regard to type of delivery and complications. Pregnancy outcomes will be compared to an age and race matched group of women who do not have Hepatitis C.

Study Hypothesis:

We expect a higher incidence of Hepatitis C in this inner city population compared to the general Canadian pregnant population (0.9%). We predict an HCV seroprevalence (rate) ranging between 2-6% in this population and we also predict that targeted screening by standardized questionnaire will fail to identify half of the Hepatitis C positive cases.

By following this group of Hepatitis C positive women through pregnancy, we expect to lend further support to previous data showing significant decrease and/or normalization of serum transaminases as well as significant increase in HCV viral load by third trimester. We also expect to see no significant differences in pregnancy outcomes or obstetrical complications between HCV positive women and the HCV negative women.

DETAILED DESCRIPTION:
All women attending our prenatal clinic will be invited to participate in this research study. Participants will complete two short questionnaires during their first visit to our prenatal clinic and be tested for Hepatitis C. Women who test positive for Hepatitis C will be carefully followed during their pregnancies and will have viral load tests and liver function tests during each trimester, at delivery and six weeks after their babies are born. All women testing positive for Hepatitis C will be referred to a hepatologist (a liver specialist) after delivery and their babies will be referred to a pediatrician for further follow-up and care. Based on previous studies we are concerned that some women may never know that they are carriers unless their blood is checked for the virus. Currently testing for Hepatitis C during pregnancy is not routinely done.

The results of this study will help us to find out how many women attending our prenatal clinic test positive for Hepatitis C and how many cases would have been missed if we only relied on one of the questionnaires to decide whether to do the blood test or not. (The questionnaire deals with factors that could put a person at risk for acquiring Hepatitis C). By following our Hepatitis C positive pregnant patients throughout their pregnancies, deliveries and after their babies are born we will learn more about how the virus changes during pregnancy. The type of deliveries, any complications and the overall state of health of the Hepatitis C positive mothers participating in this study will be reported. We will also be able to report on the number of babies who are born with the virus and the state of their health up to six months of age.

ELIGIBILITY:
Inclusion Criteria:

* Females are 16 years of age and over who present to the inner city health clinic for antenatal care who give their informed consent to participate in this study.
* Participants read and understand English or assisted by an interpreter / family member enabling fully informed consent and participation in this study

Exclusion Criteria:

* Females under the age of 16.
* Participants who do not read and understand English for whom no interpreters are available.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Females are 16 years of age and over who present to the inner city health clinic for antenatal care who give their informed consent to participate in this study.
Sampling Method: Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2005-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Yudin, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital - Women's Health Care Centre, Toronto, Ontario, Canada